CLINICAL TRIAL: NCT00433953
Title: Pharmacogenetics of Mycophenolic Acid in Kidney Transplant Patients
Brief Title: Genetic Drug Study of Mycophenolic Acid (CellCept) in Pediatric Kidney Transplant Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: No longer following patient and no plans to publish.
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-06-44
Record Dates: First submitted 2007-02-08; First posted 2007-02-12 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Kidney Transplant
Keywords: Pediatric Kidney Transplant; Kidney Transplant; CellCept; Mycophenolate Mofetil; Mycophenolic Acid
MeSH Terms: interventions — Mycophenolic Acid; Blood Specimen Collection

INTERVENTIONS:
Drug: Mycophenolate Mofetil (CellCept)
Behavioral: Dietary Monitoring
Behavioral: Drug Diary
Procedure: Blood Sampling

SUMMARY:
The purpose of this study is to determine how genes influence the response to mycophenolate mofetil (CellCept) in children who have had a kidney transplant. The study will look at how differences in some genes effect blood levels of mycophenolate mofetil over time in children, how often side effects occur and the way that children respond to mycophenolate mofetil.

The results may lead to better dosing based on individual needs.

DETAILED DESCRIPTION:
This is an open label, inpatient-outpatient prospective observational study to determine whether the inter-patient variability in mycophenolic acid (MPA) pharmacokinetics and exposure, adverse events and clinical response in pediatric transplant patients (ages 2-18 years) is associated with identifiable pharmacogenetic factors. Specific aims: 1.) To determine whether common polymorphic variations in the uridine diphosphate-glucuronosyltransferases (UGTs) are associated with inter-individual variability in MPA pharmacokinetics and exposure (by affecting MPA metabolism). 2.) To determine whether common polymorphic variations in the uridine diphosphate-glucuronosyltransferases (UGTs) are associated with inter-patient differences in the incidence of adverse events (by affecting the formation of the acyl-glucuronide metabolite). Enrolled subjects will have been receiving mycophenolate mofetil as part of their clinical standard of care. It is anticipated that the clinical portion of the study will last up to 4 hours at one study visit to include one pharmacogenetic blood sample and 4 pharmacokinetic blood samples collected out to 3 hours post-dose. Safety data to be collected will include standard of care physical exam and safety laboratory tests as well as data on adverse events and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects and non-pregnant female subjects aged 2 to 18 years who are about to receive a kidney transplant and will be on post transplant MMF containing immunosuppressive therapy.
* A signed and dated institutional review board (IRB) approved parental/guardian informed consent form and an IRB approved child assent form if applicable.
* Subjects with stable kidney allografts who are on a stable regimen of MMF (with tacrolimus and steroids)
* May have clinically important abnormalities on clinical and /or laboratory evaluations, only as these abnormalities relate to an underlying condition as determined by the principal investigator.

Exclusion Criteria:

* Children receiving cyclosporine therapy that may interact with MPA entero-hepatic recycling.
* Any medical condition(active or chronic) or prior surgery that may interfere with the pharmacokinetics of MMF as determined by the principal investigator.
* Concomitant medication that may interfere with the pharmacokinetics of MMF as determined by the principal investigator.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2007-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The following outcome measures will be performed at the study visit after the patient is on a steady state dose of mycophenolate mofetil: | Day 1
Drug measurement of MPA, MPA-G and acyl-MPA-G | Day 1
Genomic DNA extraction using standard procedures. Patients will be genotyped for the UGT2B7, UGT1A8, UGT1A9 polymorphism. | Day 1

SECONDARY OUTCOMES:
Concomitant medications and mycophenolate mofetil drug diary | Day 1
Physical Exam | Day 1
Safety Laboratory tests | Day 1
Dietary Monitoring | Day 1
Adverse Event Reporting | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Alexander A. Vinks, Pharm.D., Ph.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States